CLINICAL TRIAL: NCT04546828
Title: A Single-arm Study of Gemcitabine, Cisplatin, and Nab-Paclitaxel as Neoadjuvant Therapy for Resectable Oncologically High-Risk Intrahepatic Cholangiocarcinoma in Korea
Brief Title: A Single-arm Study of Gemcitabine, Cisplatin, and Nab-Paclitaxel as Neoadjuvant Therapy for Resectable Oncologically High-Risk IHCC in Korea
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: problem of sponsor
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Joon Oh Park, Principal Investigator, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-05-007
Record Dates: First submitted 2020-09-04; First posted 2020-09-14 (Actual); Last update posted 2022-06-15 (Actual); Status verified 2022-06

CONDITIONS: Intrahepatic Cholangiocarcinoma
MeSH Terms: conditions — Cholangiocarcinoma | interventions — Gemcitabine; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Gemcitabine, Cisplatin, and Nab-Paclitaxel (Experimental): * Nab-paclitaxel 100mg/m2 in NS dilute to a total concentration of 5 mg/mL (DO NOT FILTER) over 30 minute IV infusion on days 1 and 8 repeated every 21 days, followed by:
  * Cisplatin 25mg/m2 in 500 mL of NS over 60 minute IV infusion on days 1 and 8 repeated every 21 days, followed by:
  * Gemcitabine 800 mg/m2 in 500ml over 30 minute IV infusion on days 1 and 8 repeated every 21 days
  Interventions: Drug: Gemcitabine, Cisplatin, and Nab-Paclitaxe

INTERVENTIONS:
Drug: Gemcitabine, Cisplatin, and Nab-Paclitaxe — * Nab-paclitaxel 100mg/m2 in NS dilute to a total concentration of 5 mg/mL (DO NOT FILTER) over 30 minute IV infusion on days 1 and 8 repeated every 21 days, followed by:
  * Cisplatin 25mg/m2 in 500 mL of NS over 60 minute IV infusion on days 1 and 8 repeated every 21 days, followed by:
  * Gemcitabine 800 mg/m2 in 500ml over 30 minute IV infusion on days 1 and 8 repeated every 21 days .

SUMMARY:
1. Phase of Development: II
2. Patient Population: Resectable Oncologically High-Risk Intrahepatic Cholangiocarcinoma
3. Estimated Number of Patients: 34 patients
4. Primary Objective: To assess the resetability of neoadjuvant chemotherapy including gemcitabine, cisplatin, and nab-paclitaxel for resectable oncologically high-risk intrahepatic cholangiocarcinoma that is treated with surgical resection. Thus, the primary aim is to increase R0 resection rate via completion of all treatment
5. Secondary Objectives:

1) To assess the radiological response rate according to Response Evaluation Criteria in Solid Tumors (RECIST) 2) To determine the overall resection rate 3) To determine recurrence-free survival (RFS) 4) To identify patients' overall survival (OS) rate. 5) Saftey and tolerability 6.Exploratory Endpoint : QoL analysis via EORTC QLO C-30

DETAILED DESCRIPTION:
This is a multi-institution, open label phase II study designed to investigate the feasibility of gemcitabine/cisplatin/nab-paclitaxel as a neoadjuvant systemic chemotherapy for patients with reseactable oncologically high-risk IHCCA. This study will enroll up to 34 patients from all participating institutions with an accrual rate of 2 patients per month.

This will be an open-label, single arm study with each cycle equal to 21 days. All three drugs will be administered intravenously on day 1 and day 8 of each cycle. Dosing will be calculated using body surface area (BSA) based on the actual weight of the patient at each visit. Nab-Paclitaxel will be given at 100 mg/m2, followed by cisplatin at 25 mg/m2 and then gemcitabine at 800 mg/m2 for 2 weeks in a row followed by a week of rest. Patients will receive 4 cycles of neoadjuvant systemic chemotherapy. Restaging will be done after every 2 cycles (+/- 1 week) by radiological imaging. If radiological scans demonstrate stable disease or partial or complete tumor response and the tumor remains resectable, surgery will be performed. For patients with radiological scans that document disease progression during the study, treatment will be discontinued off the protocol and will not be evaluable for other secondary endpoints. Resection will be performed per standard of care and will include a portal lymphadenectomy for all cases. Objective evidence of recurrent disease after resection will be recorded at the time of recurrence. Patients will be followed for overall survival endpoint as well.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of intrahepatic cholangiocarcinoma
2. Oncologic high-risk disease at the time of enrollment defined as T-stage ≥ Ib (Ib - IV) Solitary lesion > 5 cm
3. Multifocal tumors or satellite lesions present confined to the same lobe of the liver as the dominant lesion but still technically resectable
4. Presence of major vascular invasion but still technically resectable
5. Suspicious or involved regional lymph nodes (N1)
6. No distant extrahepatic disease (M0)
7. High-quality cross-sectional imaging (CT or MRI) performed within 4 weeks prior to enrollment
8. Adults >18 years of age
9. Able to give informed consent
10. Able to adhere to study visit schedule and other protocol requirements
11. ECOG performance status of 0-1
12. Absolute neutrophil count ≥ 1500/mm3 13Platelet count ≥ 100,000/mm3

14.Albumin ≥3 g/dl

Exclusion Criteria:

* Serum creatinine > 1.5x upper limit of normal
* Serum total bilirubin > 1.5x upper limit of normal
* Presence of active infection
* Pregnant and/or breastfeeding
* Active other primary malignancy
* Concurrent severe and/or uncontrolled medication conditions which could compromise participation in study such as unstable angina, MI within 6 months, unstable symptomatic arrhythmia, symptomatic CHF, serious active or uncontrolled infection after inadequate biliary drainage if tumor obstructing bile duct.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-02-01 (Estimated); Primary Completion 2021-08-18 (Actual); Study Completion 2021-08-18 (Actual)

PRIMARY OUTCOMES:
Increased rate of RO resection | 16weeks

SECONDARY OUTCOMES:
the radiological response rate | 8weeks
  To assess the radiological response rate according to Response Evaluation Criteria in Solid Tumors